CLINICAL TRIAL: NCT03434210
Title: The Effect of a Community-based Long-acting Antipsychotic-treated Management Model on the Violence Risk of Patients With Schizophrenia: a 49 Weeks, Open-label Cluster Randomized Controlled Study
Brief Title: The Effect of a Community-based LAT-treated Management Model on the Violence Risk of Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yi Li MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Yi Li MD, PhD, Research clinician, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WG17A002
Record Dates: First submitted 2018-02-02; First posted 2018-02-15 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia; violence risk; long-acting antipsychotics; community-based
MeSH Terms: conditions — Schizophrenia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor would not known the arm, and forbiden to ask and comminicate with patients about the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAT-treated Community Model (Experimental): The subjects in experimental group are on 'LAT-treated Community Model'. which means,beside care as usual, subjects will be treated by paliperidone palmitate, Psychiatrists will guide community mental health professinals about the treatment and management. Psychiatrists will give community mental health professinals and patients/ caregiver long acting injection related education information.
  Interventions: Other: LAT-treated Community Model
- Care as usual (Other): The subjects in control group are on " cared as usual" Which means Patients will be managed follow the request of National Continuing Management and Intervention Program for Psychoses. Patients will managed by community mental health professionals, get education information and rehablitation guidence from them.
  Interventions: Other: care as usual

INTERVENTIONS:
Other: LAT-treated Community Model — The subjects in experimental group is on 'LAT-treated Community Model'. which means,beside care as usual, subjects will be treated by paliperidone palmitate, Psychiatrists will guide community mental health professinals about the treatment and management. Psychiatrists will give community mental health professinals and patients/ caregiver long acting injection related education information.
  Arms: LAT-treated Community Model
Other: care as usual — Control group will get usual community care, the treatment is identified by doctors, patients and care-giver as usual.
  Other Names: Control group
  Arms: Care as usual

SUMMARY:
This is a 49 weeks open-label randomized controlled study. Patients with schizophrenia and violence risk will be enrolled in the study. A community-based long-acting antipsychotics-treated management model will be applied to the experimental group, which means that professional psychiatrists will provide guidance to primary-level mental health workers on the psychotic treatment, and monthly-injected long-acting antipsychotic, paliperidone palmitate, will be used in the schizophrenia treatment. Subjects in control group will be treated and cared as usual.

DETAILED DESCRIPTION:
This is a 49 weeks open-label,cluster randomized controlled study. Patients with schizophrenia and violence risk under the government supervision will be enrolled in the study. A community-based long-acting antipsychotics-treated management model will be applied to the experimental group, which means that professional psychiatrists will provide guidance to primary-level mental health workers on the psychotic treatment, and monthly-injected long-acting antipsychotic, paliperidone palmitate, will be used in the schizophrenia treatment. The subjects in experimental group will be injected with 150mg eq and 100mg eq paliperidone palmitate in the deltoid at the 1st and 8th day, and afterwards a flexible dose of paliperidone palmitate from 75 to 150mg eq will be administrated monthly per clinical judgement. For subjects who did not take risperidone, paliperidone extended release tablets, risperidone microspheres or paliperidone palmitate for injection previously, subjects should take oral paliperidone or risperidone sustained release tablets in the screening phase to perform ultra-sensitive test (the minimum dose of risperidone 1 mg/day and the minimum dose of sustained-release tablets paliperidone 3 mg/day, at least orally three days). Only subjects who were judged by the treating physician as tolerance to the drug could usepaliperidone palmitate .Suggest previous antipsychotics could be withdrawn within 4 weeks after first paliperidone palmitate administration , but will follow doctors' clinical judgement. The study protocol does not limit other medication or treatment measures except the injectable paliperidone palmitate. Other medication or treatment measures should be decided by doctors' clinical judgement and align with patients and caregivers.Subjects in control group will be treated and cared as usual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders , Fifth Edition (DSM-V)
* Had violent behavior such as smashing or breaking, threatening with a weapon, committing arson or explosion in the past one year, whether the behavior can be stopped by persuading or not;
* Living with a guardian or a caregiver;
* Informed consent from the patients or their guardians;
* Resulted negative in urine pregnancy test if female at their reproductive age; female subjects must take effective measures to prevent pregnancy during the whole study or have been postmenopausal.-

Exclusion Criteria:

* Patients who have had suicidal ideation or suicidal attempts within 12 months before screening or in screening period;
* Intravenous drug abuse or Opioid dependence within 3 months before screening;
* Patients with treatment-resistant schizophrenia;
* Large dose of Clozapine (≥200mg/day) or other long-acting injectable antipsychotics used within 3 months or within 2 drug half-life periods before screening;
* Patients with any severe or unstable cardiovascular, respiratory, nervous system or other system diseases; clinically significant abnormality in laboratory examinations or ECG;
* Communication difficulties caused by cognitive impairment or unable to complete the assessments in the study;
* Patients assessed as unsuitable for the study in other reasons, such as allergic or intolerant to risperidone or paliperidone, resistant to risperidone or paliperidone (ineffective after adequate dosage and duration in medical history); unable to provide informed consent; historical treatments which might effect the results of the study; historical neuroleptic malignant syndrome or tardive dyskinesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-05-05 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Violence Risk Assessment For Psychiatric Patients | 49 Weeks
  The percentage of subjects rated as no or low risk (scored 0 or 1) in Violence Risk Assessment For Severe Psychiatric Patients during 49 weeks treatment
Modified Overt Aggression Scale (MOAS) | 49 Weeks
  Score change of Modified Overt Aggression Scale (MOAS ). MOAS is used to assess aggressive behavior of psychosis patients. Including Verbal aggressive, aggressive to property, aggressive to self, aggressive to others, and total score. Each domain with score 0 to 4, total weighted score 0 to 40

SECONDARY OUTCOMES:
Health economic evaluation | 49 Weeks
  Self developed health economic questionnaire, including demography questions, income before and after schizophrenia onset, schizophrenia related direct and indirect cost
Positive and Negative Syndrome Scale (PANSS) | 49 Weeks
  PANSS score change. PANSS was used to assess schizophrenia psychopathology symptoms of subjects. PANSS gave a total score (total score of 30 items) and three subscale scores, positive subscale (7 items), negative subscale (7 items), general psychopathology symptoms subscale (16 items) . Each scale rated from 1 (none) to 7 (very heavy).
Hospitalization frequency | 49 Weeks
  Hospitalization due to schizophrenia during 49 weeks
WHO Quality of Life-BREF (WHOQOL-BREF) of patients | 49 Weeks
  The patients' WHOQOL-BREF score. The WHOQOL-BREF offers a short, generic, subjective quality of life (QoL) measure, 26 important questions are scored in environmental, social, physical and psychological domains, each question from 1-5.
WHO Quality of Life-BREF (WHOQOL-BREF) of caregiver | 49 Weeks
  The caregivers' WHOQOL-BREF score. WHOQOL-BREF offers a short, generic, subjective quality of life (QoL) measure, 26 important questions are scored in environmental, social, physical and psychological domains, each question from 1-5.
Visual Analogue Scale-100 (VAS 100) of patients treatment satisfication | 49 weeks
  The patients' VAS 100 score change. Patients rate according to their treatment satisfication, score from 1( extremely unsatisfied) to 100( extremely satisfied.
Visual Analogue Scale-100 (VAS 100) of caregiver's treatment satisfication | 49 weeks
  The caregivers' VAS 100 score change.Caregivers rate according to their treatment satisfication, score from 1( extremely unsatisfied) to 100( extremely satisfied.
Family Burden Scale of Diseases (FBS) | 49 Weeks
  Family burden of the patient's family. Including 26 items, score 0( no burden) to 2(heavy burden). Refer to family economy, family daily activities, family entertainment activities, family relationships, family member physical health and mental health.
Personal and Social Performance Scale (PSP) | 49 Weeks
  PSP was a clinical scoring tool that was used for personal and social function assessment in schizophrenia subjects, and the score ranged between 1 and 100. The scale defined a continuous functional status, from overall function impaired (completely lack of independent basic functions, survival is significantly dangerous) to function well. The scale takes four functional dimensions into account: a) social useful activities, including work and study, b) the relationship between the individual and society, c) self-care, and d) disturbing and aggression
Treatment Emergent Symptom Scale (TESS) | 49 Weeks
  Treatment Emergent Symptom Scale (TESS) is a checklist including common adverse event in psychotic treatment. each item rate from 0( no) to 4 (heavy)
Clinical laboratory examination | 49 weeks
  Blood routine examination
Electrocardiogram (ECG) | 49 Weeks
  ECG testing should be performed in a quiet non-interference (such as TV, mobile) environment for the subjects. Before testing ECG the subjects should rest in the supine position for at least 5 minutes and should be limited to conversation or physical activity. Twelve-lead ECG was recorded by 25 mm/sec paper speed, measuring RR, PR, QRS and QT intervals.
Adverse events | 49 weeks
  The frequency of adverse events in the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Yi Li, Doctor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan mental health center, Wuhan, Wuhan, China